CLINICAL TRIAL: NCT05722249
Title: Interventions to Promote Well-being of Nightshift Nursing Team Members
Acronym: HSWellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ChildrensNRI
Record Dates: First submitted 2023-01-11; First posted 2023-02-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Professional Quality of Life
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: The cluster randomized crossover design is selected for logistical and ethical reasons: first, we seek generalizable findings; second, randomizing individual members of the nightshift will inevitably contribute to cross-contamination of the intervention arms; having a control group will similarly be at risk of contamination from peers randomly assigned to intervention arms as nightshift workers are assigned to float to other units when staffing needs merit such assignments; and given the known potential health risks for some nightshift workers, not providing an intervention could be considered unethical. In the cluster cross-over design, the staff in the participating clinical inpatient units will each receive an intervention during each of two time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A, Study Period 1 (Mindfulness and Sleep Hygiene): (Experimental): Immediately after the sleep hygiene content, the overview of the mindfulness intervention will be offered. All enrolled participants in Arm A, Study Period 1, will attend a 15 minute in-person "Introduction to Mindfulness" session after randomization.
  Interventions: Behavioral: Mindfulness and Sleep Hygiene
- Arm B, Study Period 1 (Physical Activity and Sleep Hygiene): (Active Comparator): All enrolled participants in the inpatient units randomly assigned to Arm B during Study Period 1 will receive written guidelines about physical activity during the nightshift (please see Appendix V). These guidelines will instruct them to achieve the goal of up to 15 minutes of physical activity between midnight and 0500 each nightshift during the 8-week study period. Each enrolled participant will view a video with voice over of the study team physical therapist demonstrating the methods.
  Interventions: Behavioral: Phyical activity and Sleep Hygiene

INTERVENTIONS:
Behavioral: Mindfulness and Sleep Hygiene — Participants will experience demonstrations and explanations regarding sleep hygiene, mindfulness alerts for at work and mindfulness rest for at home.
  Arms: Arm A, Study Period 1 (Mindfulness and Sleep Hygiene):
Behavioral: Phyical activity and Sleep Hygiene — All enrolled participants in the inpatient units randomly assigned to Arm B during Study Period 1 will receive written guidelines about physical activity during the nightshift (please see Appendix V). These guidelines will instruct them to achieve the goal of up to 15 minutes of physical activity between midnight and 0500 each nightshift during the 8-week study period. Each enrolled participant will view a video with voice over of the study team physical therapist demonstrating the methods
  Arms: Arm B, Study Period 1 (Physical Activity and Sleep Hygiene):

SUMMARY:
Background:

Nightshift health care employees can experience greater likelihood of health threats such as weight gain, hypertension, and sleep disturbances. Evidence indicates a willingness of nightshift health care professionals to engage in wellness activities initiated at the work setting and during the assigned nightshift. In this single site study at a freestanding pediatric tertiary care hospital, inpatient units will be randomized to one of two nightshift interventions during an 8-week study period (mindfulness plus sleep hygiene or physical activity plus sleep hygiene). Immediately following the first study period, the randomized units will begin a second study period in which they will continue with the intervention first received but shall add the intervention not initially received. While there are hundreds of studies that describe the adverse health and safety effects of night shift work, there are few studies where interventions are tested for their efficacy to reduce the harm to workers or improve their well-being. Currently the few intervention studies that exist focus on the scheduling, duration and timing of work shifts, the timing of meals, and aspects of lighting in the workplace. Other interventions, such as those proposed in this study, have not been tested systematically using a rigorous design.

Purpose and Methods:

The purpose of this study, using a cluster cross-over randomized trial design, is to measure the impact on professional quality of life (primary endpoint) and medication administration error, role-related meaning, and sleep quality (secondary endpoints) of either a mindfulness intervention plus sleep hygiene (Arm A) or a physical activity intervention plus sleep hygiene (Arm B) in the first study period, and the combination of both interventions on the same outcomes in the second study period for nightshift health care employees.

DETAILED DESCRIPTION:
Study Purpose The purpose of this study, using a cluster cross-over randomized trial design involving inpatient units at a freestanding pediatric hospital, is to measure the impact on professional quality of life (primary endpoint), medication administration error, role-related meaning, and sleep quality (secondary endpoints) of either a mindfulness intervention (Arm A) or a physical activity intervention (Arm B) in the first study period, and the combination of both interventions on the same outcomes in the second study period for nightshift health care employees.

Primary Objective

1.The primary objective of this study is to determine and compare the impact on professional quality of life (as measured by the ProQOL scale) of either a mindfulness intervention (Arm A) or a physical activity intervention (Arm B) during an 8-week study period (study period 1).

1h1: ProQOL scale mean scores for compassion satisfaction will increase in both study arms during study period 1 from baseline (the week prior to randomization to the study Arms) to the end of the 8-week study period (Week 8).

1h2: ProQOL scale mean scores for compassion fatigue will decrease in both study arms during study period 1 from baseline (the week prior to randomization to the study Arms) to the end of the 8-week study period (Week 8).

1h3: ProQOL scale mean scores for compassion satisfaction will not differ at baseline (the week prior to randomization to the study Arms) or at the end of the first study period (Week 8) between the two study arms.

1. h4. ProQOL mean scores for compassion fatigue will not differ between the two arms at baseline (the week prior to randomization to the study Arms) or at the end of the first study period (Week 8).

   Secondary Objectives 2. Determine and compare the impact on professional quality of life (as measured by the ProQOL scale) of the combined mindfulness intervention and physical activity intervention (Arms A and B) during a second 8-week study period (study period 2) as compared to the first study period.
2. h1: ProQOL scale mean scores for compassion satisfaction will increase in both study arms during study period 2 from the end of the first 8-week study period (Week 8) to the end of the second study period (Week 16), and from baseline to Week 16.

2h2: ProQOL scale mean scores for compassion fatigue will decrease in both study arms during study period 2 from the end of the first 8-week study period (Week 8) to the end of the second study period (Week 16), and from baseline to Week 16.

2h3: ProQOL scale mean scores for compassion fatigue will not differ between the two arms at Week 8 or at the end of the second study period (Week 16).

2h4. ProQOL scale mean scores for compassion satisfaction will not differ between the two arms at Week 8 or at the end of the second study period (Week 16).

3. Determine and compare the impact of the interventions by study period on role-related meaning as measured by the Role-Related Meaning Scale (RRMS) and sleep quality as measured by the PROMIS Sleep Disturbance measure and the PROMIS Sleep-Related Impairment Measure (SRI).

3h1: the RRMS mean scores will increase and PROMIS Sleep Disturbance and SRI mean scores will decrease in both study arms from baseline to Week 8, from Week 8 to Week 16, and from baseline to Week 16.

3h2: the RRMS mean scores and the PROMIS Sleep Disturbance and SRI mean scores will not differ between the two arms at baseline, Week 8 or at Week 16.

4. Determine the impact of the intervention periods (Week 8, Week 16) on a patient-related indicator, Medication Administration Error as compared to the error rate at baseline.

4h1: Medication Administration Errors will not differ between the two study arms at baseline, Week 8 or at Week 16.

4h2: Medication Administration Errors will decrease within both study arms from baseline to Week8, and from Week 8 to Week 16.

General Design Description The study design is a cluster cross-over randomized trial involving 11 inpatient units at a freestanding pediatric hospital. In the randomization, the 11 units will be randomized to two study arms (Arm A - mindfulness intervention plus sleep hygiene information; Arm B - physical activity plus sleep hygiene information) during the first 8-week study period. Immediately following this study period, the units assigned to each arm will cross and receive the intervention not received in the first study period plus the ongoing access to the previous intervention. Both arms in the first study period will have education content specific to sleep hygiene connected to the existing napping option.

The cluster randomized crossover design is selected for logistical and ethical reasons: first, we seek generalizable findings; second, randomizing individual members of the nightshift will inevitably contribute to cross-contamination of the intervention arms; having a control group will similarly be at risk of contamination from peers randomly assigned to intervention arms as nightshift workers are assigned to float to other units when staffing needs merit such assignments; and given the known potential health risks for some nightshift workers, not providing an intervention could be considered unethical. In the cluster cross-over design, the staff in the participating clinical inpatient units will each receive an intervention during each of two time periods. Interventions, such as physical activity and mindfulness, that can be done at the group level and may be more effective when done with a group, are ideal for this design (Arnup et al., 2014; Arnup et al., 2017; Parienti & Kuss, 2007; Moerbeek, 2020; Reich et al., 2012). This design is also selected for its efficiency and reduced costs compared with a clinical trial with individuals being randomized (Taljaard et al, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be nurses and members of the nursing care team that work the nightshift fulltime or that rotate from the dayshift to the nightshift on a routine basis. Participants will need to be scheduled to work at least 2 weeks of the nightshift during each study period (Study Period 1, Study Period 2) to be fully eligible to participate in the study. To be fully eligible, participants must be able to complete a consent process and understand the study design and the self-report periods.

Exclusion Criteria:

* Exclusion criteria would include nurses and nursing care team members who do not rotate regularly to the nightshift or who work only the dayshift.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Professional Quality of Life Scale, (ProQOL-21). The primary outcome variable will be change in professional quality of life as measured by the Professional Quality of Life Scale, (ProQOL-21). | baseline or the week before randomization, Week 8 and Week 16
  The ProQOL contains two domains: Compassion Satisfaction and Compassion Fatigue. For this study, we shall administer the ProQOL-21, a revised version of the ProQOL derived from a Rasch analysis (Heritage, et al., 2018) where higher scores mean better professional quality of life.

SECONDARY OUTCOMES:
change in Role-Related Meaning | Baseline or the week before randomization, Week 8 and Week 16
  Role-Related Meaning Scale (RRMS): Role-related meaning is defined as internalized, individualized awareness of personal values, and the extent to which these values are concordant with those of the role, work setting or work culture. In this study, role-related meaning will be measured using the Role-related Meaning Scale for Staff (RRMS) where higher scores mean better role meaning.

OTHER OUTCOMES:
Change in the PROMIS Sleep Disturbance Measure | Baseline or the week before randomization, Week 8 and Week 16
  PROMIS Sleep Disturbance Measure: The 8-item short-form for this measure with its 5-point Likert response format will be used in this study; higher scores mean more disturbed sleep.
Change in the PROMIS Sleep-Related Impairment Measure (SRI) | Baseline or the week before randomization, Week 8 and Week 16
  PROMIS Sleep-Related Impairment Measure (SRI): This 8-item short-form measure was similarly developed and is similarly formatted and structured as the PROMIS Sleep Disturbance; higher scores mean more impaired sleep.
Change in Medication Error Administration | 60 days before Baseline, Week 8 and Week 16
  Medication Error Administration: The exploratory outcome variable is Medication Error Administration. According to the National Coordinating Council for Medication Error Reporting and Prevention (NCCMERP) a "medication error" is defined as "any preventable event that may cause or lead to inappropriate medication use or patient harm while the medication is in the control of the healthcare professional, patient or parent; the higher number means more errors were made.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Hinds, PhD, RN, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Group summary will be provided to all upon request immediately after their publication by the study team.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The above will be made available immediately after the publication of study outcomes by the study team.
Access Criteria: A written request to the study PI will initiate the process of sharing the above items.